CLINICAL TRIAL: NCT03081741
Title: A Prospective Study of Circulating Tumor DNA Detection in Surveillance for Lung Cancer Patients
Brief Title: Circulating Tumor DNA in Surgical Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen Gene Health Bio Tech Co., Ltd. (Industry)
Collaborators: Shenzhen People's Hospital (Other); Shenzhen Second People's Hospital (Other); Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GeneHealth-LC-01
Record Dates: First submitted 2017-03-12; First posted 2017-03-16 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and FFPE tissue sections were collected from each patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Conduct a prospective study to detect the change of ctDNA of surgical lung cancer patients.

DETAILED DESCRIPTION:
Studies have shown the feasibility of detecting mutation status by blood circulating tumor DNA (ctDNA) in lung cancer patients.

The investigators plan to test the blood ctDNA in surveillance of surgical lung cancer patients. And evaluate the correlation between ctDNA level with tumor relapse or metastasis.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 to 80 years Undergo radical surgery Histologically confirmed diagnosis of lung cancer Considered primary lung cancer by clinical criteria Patients must have given written informed consent

Exclusion Criteria:

Unable to comply with the study procedure Malignant tumor history Patients who received any treatment prior to resection Unqualified blood samples

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical lung cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2020-03-18 (Estimated)

PRIMARY OUTCOMES:
Effect of surgery on ctDNA of lung cancer patients | before surgery and 7days after surgery
  Changes of blood ctDNA of lung cancer patients before and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Geng Tian, MD, Study Chair — Shenzhen Second People's Hospital
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng M, Xie Y, Li X, Qian Y, Tu X, Yao X, Cheng F, Xu F, Kong D, He B, Liu C, Cao F, Yang H, Yu F, Xu C, Tian G. Resectable lung lesions malignancy assessment and cancer detection by ultra-deep sequencing of targeted gene mutations in plasma cell-free DNA. J Med Genet. 2019 Oct;56(10):647-653. doi: 10.1136/jmedgenet-2018-105825. Epub 2019 Apr 13. PMID 30981987